CLINICAL TRIAL: NCT01852292
Title: Double Blind, Placebo Controlled Study Assessing the Efficacy of Buparlisib (BKM120) Plus Paclitaxel Versus Placebo Plus Paclitaxel in Patients With Platinum Pre-treated Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Study of Efficacy and Safety of Buparlisib (BKM120) Plus Paclitaxel Versus Placebo Plus Paclitaxel in Recurrent or Metastatic Head and Neck Cancer Previously Pre-treated With a Platinum Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBKM120H2201; 2013-000744-26 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: platinum pre-treated recurrent or metastatic; Head and neck squamous cell carcinoma; recurrent; metastatic; BKM120
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Recurrence | interventions — NVP-BKM120; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buparlisib + weekly Paclitaxel (Experimental): Patients who were randomized to this arm on a 1:1 randomization, took buparlisib 100 mg daily and paclitaxel 80 mg/m^2 weekly.
  Interventions: Drug: Buparlisib; Drug: Paclitaxel
- Buparlisib matching placebo + Paclitaxel (Placebo Comparator): Patients who were randomized to this arm on a 1:1 randomization, took buparlisib matching placebo 100 mg daily and paclitaxel 80 mg/m^2 weekly.
  Interventions: Drug: Buparlisib matching Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: Buparlisib — Buparlisib comes in gelatin capsules and is taken orally at a dose of 100 mg/day.
  Other Names: BKM120
  Arms: Buparlisib + weekly Paclitaxel
Drug: Buparlisib matching Placebo — Buparlisib matching placebo comes in gelatin capsules and is taken orally at a dose of 100 mg/day.
  Arms: Buparlisib matching placebo + Paclitaxel
Drug: Paclitaxel — Paclitaxel is an intravenous infusion that is given once every week in 80 mg/m^2.

SUMMARY:
Phase II Study of efficacy and safety of buparlisib (BKM120) plus paclitaxel versus placebo plus paclitaxel in recurrent or metastatic Head and Neck cancer previously pre-treated with a platinum therapy.The primary endpoint was PFS and the key secondary endpoint was Overall Survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically/cytologically-confirmed HNSCC.
* Patient has archival or fresh tumor tissue for the analysis of PI3K-related biomarkers. One tumor block (preferred) or a minimum of 12 unstained slides to be provided. Enrollment in the study is contingent on confirmation of an adequate amount of tumor tissue.
* Patients with recurrent or metastatic disease resistant to platinum-based chemotherapy (defined as progression while on platinum-based chemotherapy given in the recurrent/metastatic setting). Pretreatment with cetuximab is allowed
* Measurable disease as determined by per RECIST criteria v1.1. If the only site of measurable disease is a previously irradiated lesion, documented progression of disease and a 4 week period since radiotherapy completion is required
* Adequate bone marrow function and organ function
* ECOG Performance Status ≤ 1

Exclusion Criteria:

* Patient has received previous treatment with any AKT, mTOR inhibitors or PI3K pathway inhibitors;
* Patient treated with more than one prior chemotherapy regimen for recurrent/metastatic disease
* Patient has symptomatic CNS metastases. Patients with asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior local treatment for CNS metastases ≥ 28 days prior to the start of study treatment (including radiotherapy and/or surgery) and must have stable low dose of corticosteroid therapy;
* Patient has not recovered to ≤ grade 1 (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient has any of the following cardiac abnormalities:symptomatic congestive heart failure, history of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy, Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO); myocardial infarction ≤ 6 months prior to enrolment, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, symptomatic pericarditis, QTcF > 480 msec on the screening ECG (using the QTcF formula);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (52):
- United States (7):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Dana Farber Cancer Institute IRB, Boston, Massachusetts
  - Washington U School of Medicine Center for Clinical Studies SC - BKM120H2201, St Louis, Missouri
  - The Mount Sinai Hospital Dept of Oncology, New York, New York
  - University of N.C. at Chapel Hill Lineberger Comp. Cancer Ctr., Chapel Hill, North Carolina
  - University Hospitals Case Medical Center Univ. Hospitals of Cleveland, Cleveland, Ohio
  - UPMC Cancer Centers BKM120H2201, Pittsburgh, Pennsylvania
- Novartis Investigative Site, St Leonards, New South Wales, Australia
- Canada (2):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Saint-Herblain, France
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Nyíregyháza
- India (6):
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Dehli, New Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Kerala
  - Novartis Investigative Site, Mumbai
- Novartis Investigative Site, Dublin, Ireland
- Italy (7):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Venezia, VE
- Japan (3):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Koto-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
- Novartis Investigative Site, Warsaw, Poland
- Russia (3):
  - Novartis Investigative Site, Leningrad Region, Russia
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Saint Petersburg
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho-gu
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
- Taiwan (3):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Desilets A, Lucas J, Licitra LF, Lu S, Tse A, Tang T, Dreyer K, He N, Birgerson LE, Faivre S, Soulieres D. Buparlisib and Paclitaxel in Patients with Head and Neck Squamous Cell Carcinoma: Immunogenomic Biomarkers of Efficacy from the BERIL-1 Study. Target Oncol. 2025 Mar;20(2):299-310. doi: 10.1007/s11523-024-01126-0. Epub 2025 Jan 14. PMID 39808408
- [Derived] Soulieres D, Faivre S, Mesia R, Remenar E, Li SH, Karpenko A, Dechaphunkul A, Ochsenreither S, Kiss LA, Lin JC, Nagarkar R, Tamas L, Kim SB, Erfan J, Alyasova A, Kasper S, Barone C, Turri S, Chakravartty A, Chol M, Aimone P, Hirawat S, Licitra L. Buparlisib and paclitaxel in patients with platinum-pretreated recurrent or metastatic squamous cell carcinoma of the head and neck (BERIL-1): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Oncol. 2017 Mar;18(3):323-335. doi: 10.1016/S1470-2045(17)30064-5. Epub 2017 Jan 26. PMID 28131786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned: 150; Analyzed: 158. Patients were randomized to receive treatment with buparlisib 100 mg daily (n=79) or placebo (n=79) in combination with paclitaxel.
Pre-assignment Details: 158 patients randomized in a 1:1 ratio to treatment with buparlisib plus paclitaxel or placebo plus paclitaxel; stratification: number of prior lines of treatment in the recurrent/metastatic setting (1 vs.2) & region of Investigator site (North America vs. Rest of the World). In this study, Not Completed = Discontinued study treatment per Protocol
Groups:
- Buparlisib + Weekly Paclitaxel: Patients who were randomized to this arm on a 1:1 randomization, took buparlisib 100 mg daily and weekly paclitaxel.
- Buparlisib Matching Placebo + Paclitaxel: Patients who were randomized to this arm on a 1:1 randomization, took buparlisib matching placebo 100 mg daily and weekly paclitaxel.
Period: Overall Study
Arm/Group | Buparlisib + Weekly Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Started | 79 | 79
Completed | 0 (Completed = participants who were ongoing and did not discontinue study treatment per protocol) | 0 (Completed = participants who were ongoing and did not discontinue study treatment per protocol)
Not Completed | 79 | 79
Not completed — Untreated - did not receive study drug | 3 | 1
Not completed — Death | 9 | 8
Not completed — Patient/guardian decision | 8 | 4
Not completed — Adverse Event | 8 | 11
Not completed — Physician Decision | 6 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 1
Not completed — Progressive disease | 42 | 52

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Groups:
- Buparlisib + Paclitaxel: Patients who were randomized to this arm on a 1:1 randomization, took buparlisib 100 mg daily and paclitaxel 80 mg/m^2 weekly.
- Total: Total of all reporting groups
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
  Years | 58.0 (9.44) | 58.2 (9.44) | 58.1 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
  Participants
    Female | 14 | 11 | 25
    Male | 65 | 68 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
  Participants
    Hispanic or Latino | 3 | 0 | 3
    East Asian | 12 | 9 | 21
    Southeast Asian | 4 | 9 | 13
    South Asian | 6 | 5 | 11
    Russian | 7 | 4 | 11
    Mixed ethnicity | 1 | 2 | 3
    Not reported | 13 | 10 | 23
    Unknown | 3 | 6 | 9
    Other | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: PFS was defined as the time from the date of randomization to the date of the event, defined as the first radiologically documented disease progression per RECIST v. 1.1 or death due to any cause. If a patient has not progressed or died at the analysis cut-off date or when the patient receives further anti-neoplastic therapy, PFS was censored on the date of the last adequate tumor assessment before the earlier of the cut-off date or start of the further anti-neoplastic therapy date.
Time Frame: 4 weeks and thereafter every 6 weeks until disease progression or death up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
months | 4.63 [3.52 to 5.32] | 3.45 [2.17 to 3.71]
Statistical Analysis 1: Comparison: Buparlisib + Paclitaxel vs Buparlisib Matching Placebo + Paclitaxel; Test type: Other — Double Criteria for PFS; Cox Proportional Hazard = 0.646, 95% CI 2-sided [0.44 to 0.94]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut-off, OS was censored at the date of last contact.
Time Frame: 4 weeks and thereafter every 6 weeks until disease progression or death up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
months | 10.41 [7.29 to 12.78] | 6.54 [5.26 to 8.77]
Statistical Analysis 1: Comparison: Buparlisib + Paclitaxel vs Buparlisib Matching Placebo + Paclitaxel; Test type: Other — Double criteria for OS; Cox Proportional Hazard = 0.72, 95% CI 2-sided [0.49 to 1.04]

3. Secondary Outcome: Overall Response Rate (ORR) as Per Local Radiological Assessment
Description: ORR: percentage of patients with best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1. CR is defined as disappearance of all target lesions and any pathological lymph nodes must have a short axis of <10 mm and the disappearance of all non-target lesions). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters or the persistence of 1 or more non-target lesions or lymph nodes identified as a site of disease at Baseline with a short axis of ≥10mm).
Time Frame: 4 weeks and thereafter every 6 weeks until disease progression or death up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
Percentage of participants | 39.2 [28.4 to 50.9] | 13.9 [7.2 to 23.5]

4. Secondary Outcome: Time to Response (TTR) as Per Local Radiological Assessment
Description: TTR is the time from date of randomization until first documented response (CR or PR, which has to be confirmed subsequently) according to RECIST v1.1. CR is defined as disappearance of all target lesions and any pathological lymph nodes must have a short axis of <10 mm and the disappearance of all non-target lesions). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters or the persistence of 1 or more non-target lesions or lymph nodes identified as a site of disease at Baseline with a short axis of ≥10mm).
Time Frame: 4 weeks and thereafter every 6 weeks until disease progression or death up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
months | 1.02 [0.8 to 9.2] | 0.99 [0.8 to 5.1]

5. Secondary Outcome: Disease Control Rate (DCR) as Per Local Radiological Assessment
Description: DCR is the percentage of patients with a best overall response of CR, PR or stable disease (SD), according to RECIST v1.1. CR is defined as disappearance of all target lesions & any pathological lymph nodes must have a short axis of <10 mm & the disappearance of all non-target lesions). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters or the persistence of 1 or more non-target lesions or lymph nodes identified as a site of disease at Baseline with a short axis of ≥10mm). SD is defined as neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2.
Time Frame: 4 weeks and thereafter every 6 weeks until disease progression or death up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
Percentage of participants | 72.2 [60.9 to 81.7] | 69.6 [58.2 to 79.5]

6. Secondary Outcome: Duration of Response (DoR) as Per Local Investigator
Description: DoR is the time from the date of the first documented response (CR or PR, which had to be confirmed subsequently) to the date of the first radiologically documented disease progression or death due to disease according to RECIST v1.1 .
Time Frame: 4 weeks and thereafter every 6 weeks until disease progression or death up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
months | 3.06 [2.1 to 9.6] | 4.17 [2.7 to 5.6]

7. Secondary Outcome: Health-related Quality of Life (HRQoL):Time to 10% Definitive Deterioration in the Global Health Status/Quality of Life Per EORTC-QLQ-C30
Description: A summary of EORTC-QLQ-C30 scores by time window. Time to deterioration is the number of days between the date of randomization and the date of the assessment at which definitive deterioration is seen. Definitive Deterioration in global health status and symptoms was defined as a decrease in the subscale score by at least 10% compared to baseline, with no later increase above this threshold observed during the course of the study. If a patient had not had an event prior to analysis cut-off or start of another anticancer therapy, time to deterioration was censored at the date of the last quality of life (QoL) evaluation.
Time Frame: Baseline, every 6 weeks starting from cycle 2 day 15 up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
months | 3.0 [1.6 to 4.9] | 3.5 [2.1 to 4.3]

8. Secondary Outcome: Health-related Quality of Life (HRQoL):Time to 10% Definitive Deterioration in the Head and Neck Cancer Symptoms Scales for Pain, Speech Problems, Swallowing and Sense Problems Per EORTC-QLQ-HN35
Description: A summary of EORTC-QLQ-HN35 scores by time window. Time to deterioration is the number of days between the date of randomization and the date of the assessment at which definitive deterioration is seen. Definitive Deterioration in global health status and symptoms was defined as an increase in the subscale score of at least 10% compared to baseline, with no later decrease above this threshold observed during the course of the study. If a patient had not had an event prior to analysis cut-off or start of another anticancer therapy, time to deterioration was censored at the date of the last quality of life (QoL) evaluation.
Time Frame: Baseline, every 6 weeks starting from cycle 2 day 15 up to 3.5 years
Population: The Full analysis set (FAS) includes all patients who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
Number analyzed (Participants) | 79 | 79
Months
  Pain Subscale | 5.8 [4.2 to 7.3] | 5.3 [3.2 to 6.8]
  Speech problems | 5.6 [4.1 to 6.9] | 4.2 [2.2 to 5.4]
  Swallowing | 5.1 [3.7 to 7.2] | 4.6 [2.8 to 6.7]
  Sense Problems | 5.1 [3.1 to 7.3] | 4.6 [2.9 to 6.5]

9. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 Pharmacokinetics (PK) for AUC0-24 and AUClast
Description: To Characterize PK of buparlisib given in combination with paclitaxel for AUC0-24 (area under plasma concentration-time curve from time 0 to end of dosing interval of 24 hours) & AUClast (AUC from time 0 to last measurable concentration sampling time).
Time Frame: Time point(s) at which PK samples for Non-Compartmental analysis were collected were 0, 0.5,1,1.5, 2, 3, 4, 6, 9 and 24 hours at Cycle 1, Day 15
Population: Full Sampling Pharmacokinetic Analysis Set (FPAS): All pts in PAS who received planned dose of buparlisib every day for last consecutive 7 days before full PK profile assessment on C1D15, didn't vomit within 4 hours of buparlisib dosing, had at least 1 dose of paclitaxel before collection of PK sample for PK profile & had evaluable full PK profile
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Buparlisib + Paclitaxel
Number analyzed (Participants) | 79
ng*hr/mL
  AUC0-24 (n = 4): number analyzed (Participants) | 4
  AUC0-24 (n = 4) | 25628.56 [13651.75 to 33375.10]
  AUClast (n = 4): number analyzed (Participants) | 4
  AUClast (n = 4) | 25734.33 [13651.75 to 33306.37]

10. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 Pharmacokinetics (PK) for Cmax
Description: To characterize the pharmacokinetics of buparlisib given in combination with paclitaxel for Cmax.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Buparlisib + Paclitaxel
Number analyzed (Participants) | 79
ng/mL | 1775.00 [834.00 to 2180.00]

11. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 Pharmacokinetics (PK) for Tmax
Description: To characterize the pharmacokinetics of buparlisib given in combination with paclitaxel for Tmax.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Buparlisib + Paclitaxel
Number analyzed (Participants) | 79
hour (hr) | 2.42 [1.00 to 4.00]

12. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 Pharmacokinetics (PK) for CL/F
Description: To characterize the pharmacokinetics of buparlisib given in combination with paclitaxel for CL/F.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: L/hr
Arm/Group | Buparlisib + Paclitaxel
Number analyzed (Participants) | 79
L/hr | 4.14 [3.00 to 7.33]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 3.5 years.
Description: AEs, SAEs based on Safety Set: all pts who received at least 1 dose of study trtmnt & had at least 1 post-baseline safety assessment. Pts analyzed according to study trtmnt actually received, defined as trtmnt pt received on 1st day of study trtmnt
Arm/Group | Buparlisib + Paclitaxel | Buparlisib Matching Placebo + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 16/76 | 17/78
Serious Adverse Events (participants affected / at risk) | 43/76 | 37/78
Other Adverse Events (participants affected / at risk) | 76/76 | 75/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib + Paclitaxel (N=76) | Buparlisib Matching Placebo + Paclitaxel (N=78)
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Blindness (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Aorto-oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral cavity fistula (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 2
Face oedema (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 4
General physical health deterioration (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 2
Candida sepsis (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 6 | 6
Post procedural infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Device connection issue (Product Issues) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial rupture (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib + Paclitaxel (N=76) | Buparlisib Matching Placebo + Paclitaxel (N=78)
Anaemia (Blood and lymphatic system disorders) | 29 | 32
Leukopenia (Blood and lymphatic system disorders) | 7 | 13
Neutropenia (Blood and lymphatic system disorders) | 23 | 10
Abdominal pain (Gastrointestinal disorders) | 7 | 2
Constipation (Gastrointestinal disorders) | 14 | 8
Diarrhoea (Gastrointestinal disorders) | 26 | 13
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 9 | 5
Nausea (Gastrointestinal disorders) | 19 | 13
Odynophagia (Gastrointestinal disorders) | 4 | 1
Oral pain (Gastrointestinal disorders) | 4 | 1
Stomatitis (Gastrointestinal disorders) | 23 | 10
Vomiting (Gastrointestinal disorders) | 19 | 11
Asthenia (General disorders) | 20 | 15
Face oedema (General disorders) | 2 | 4
Fatigue (General disorders) | 31 | 16
Non-cardiac chest pain (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 5 | 10
Pyrexia (General disorders) | 12 | 16
Nasopharyngitis (Infections and infestations) | 4 | 4
Pneumonia (Infections and infestations) | 2 | 6
Respiratory tract infection (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 6 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood alkaline phosphatase increased (Investigations) | 6 | 1
Blood creatinine increased (Investigations) | 4 | 1
Blood glucose increased (Investigations) | 3 | 4
Blood lactate dehydrogenase increased (Investigations) | 5 | 5
Gamma-glutamyltransferase increased (Investigations) | 8 | 7
Neutrophil count decreased (Investigations) | 5 | 4
Weight decreased (Investigations) | 19 | 9
White blood cell count decreased (Investigations) | 7 | 3
Decreased appetite (Metabolism and nutrition disorders) | 23 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 47 | 27
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 5 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Dizziness (Nervous system disorders) | 6 | 6
Dysgeusia (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 14 | 6
Neuropathy peripheral (Nervous system disorders) | 6 | 18
Paraesthesia (Nervous system disorders) | 8 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 3
Anxiety (Psychiatric disorders) | 13 | 9
Depression (Psychiatric disorders) | 13 | 7
Insomnia (Psychiatric disorders) | 10 | 6
Mood altered (Psychiatric disorders) | 4 | 5
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 15
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 2
Erythema (Skin and subcutaneous tissue disorders) | 8 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 3
Rash (Skin and subcutaneous tissue disorders) | 14 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3
Hypertension (Vascular disorders) | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT01852292/SAP_000.pdf
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT01852292/Prot_001.pdf